CLINICAL TRIAL: NCT03164980
Title: Comparison of Quality of Life (QoL) Between Trabectedin/PLD and Standard Platinum-based Therapy in Patients With Platinum Sensitive Recurrent Ovarian, Fallopian Tube and Peritoneal Cancer
Brief Title: QoL-Comparison Between Trabectedin/PLD and Pt-based Therapy in Patients With Pt-sensitive Recurrent Ovarian Cancer
Acronym: COMPASS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A total of 204 patients were planned to be randomized. Due to slow recruitment of the trial, the recruitment was prematurely terminated after randomization of the 89th patient.
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Collaborators: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other); PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOGGO S16/COMPASS
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life; Ovarian Cancer; Recurrent Ovarian Carcinoma
Keywords: Quality of life; ovarian cancer; platinum sensitive; recurrent
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): PLD followed by Trabectedin. Treatment is repeated every 3 weeks for 6 cycles or until disease progression.
  Interventions: Drug: Trabectidin (Yondelis)
- Arm B (Experimental): * Carboplatin/PLD
  * Carboplatin/Gemcitabine
  * Carboplatin/Paclitaxel Patients will be treated for 6 cycles or until PD, unacceptable toxicity or patient's wish to discontinue, whichever occurs first.
  Interventions: Drug: Trabectidin (Yondelis)

INTERVENTIONS:
Drug: Trabectidin (Yondelis) — To compare QoL in patients treated with trabectedin/PLD vs. other standard combination therapy of carboplatin/ PLD, carboplatin/ gemcitabine, or carboplatin/ paclitaxel

SUMMARY:
This is a multicenter, randomized, controlled, open-label study including patients with recurrent, platinum-sensitive, ovarian, peritoneal or fallopian tube cancer.

The main scope of the trial is to evaluate QoL during chemotherapy comparing trabectedin/PLD with other standard platinum-based chemotherapy in platinum-sensitive disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label study including patients with recurrent, platinum-sensitive, ovarian, peritoneal or fallopian tube cancer.

The main scope of the trial is to evaluate QoL during chemotherapy comparing trabectedin/PLD with other standard platinum-based chemotherapy in platinum-sensitive disease.

Patients with recurrent, platinum-sensitive, ovarian, fallopian tube and peritoneal cancer will be stratified according to surgery for relapse (R0 vs. R1/2 resection) vs. no surgery in the same setting and age (< 75 years vs. ≥ 75 years), and randomized 1:1 to receive either trabectedin/PLD (Arm A) or one of 3 platinum-based standard therapies without bevacizumab (Arm B, "other standard therapy"). In case of randomization to "other standard therapy", the investigator has the choice between carboplatin/PLD, carboplatin/gemcitabine and carboplatin/paclitaxel. Patients in both treatment arms will receive chemotherapy up for 6 cycles or until disease progression (PD), unacceptable toxicities or patient's wish to stop therapy, whichever occurs first.

ELIGIBILITY:
Inclusion criteria

1. Women aged ≥ 18 years
2. Patients with histologically confirmed diagnosis of epithelial ovarian cancer, primary peritoneal carcinoma or fallopian tube cancer who received ≥1 prior chemotherapy
3. Patients must be eligible for platin-containing therapy; Patient is defined as platin-sensitive when considered for platin-containing therapy by the investigator. The time frame from end of prior therapy until disease progression alone is not pivotal for study participation. Patients without a platin-containing regimen in the previous line who are also eligible for platin-containing regime are also appropriate for participation
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
5. Adequate baseline organ function as defined as

   * Leucocytes > 3.0 x 109/l
   * Platelet count > 100 x 109/l
   * Absolute neutrophil count (ANC) ≥1500/mm3
   * Haemoglobin ≥ 9 g/dl
   * Alkaline Phosphatase (AP) ≤ 2.5 × ULN (consider hepatic isoenzymes 5 nucleotidase or gamma glutamyl transpeptidase (GGT), if the elevation could be osseous in origin)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN
   * Creatinine-Clearance ≥ 60 ml/min (MDRD formula or Cockroft & Gault formula)
   * Serum creatinine ≤ 1.5 mg/dl
   * Creatine phosphokinase (CPK) ≤ 2.5 × ULN
   * Total bilirubin < ULN
6. Women of childbearing potential should use contraceptives or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication or be surgically sterile.
7. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 50% as determined by echocardiogram
8. Patients must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up assessments and procedures.

Exclusion criteria

1. Only malignancies, which influence the prognosis
2. Any unstable or serious concurrent condition (e.g. active infection requiring systemic therapy).
3. Chemotherapy or radiation therapy or tumor embolization within 2 weeks prior to the first dose of study drug or planned during study participation.
4. Patients who have refractory disease. Refractory disease is defined if relapse occurs <4 months after beginning of platin-containing therapy.
5. Hypersensitivity to the active substance or to any of the excipients of study drug
6. Findings from ECG and/or assessment of LVEF which indicate an anthracycline-related cardiotoxic process which contradicts administration of liposomal doxorubicin in accordance with the requirements of the SmPC of PLD.
7. Biological therapy, immunotherapy, hormonal therapy or treatment with an investigational agent within 14 days (for bevacizumab, 30 days) prior to the first dose of study drug.
8. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
9. Participation in another clinical study with experimental therapy within the 30 days before start of and during treatment. Participation in a non-interventional study should be discussed with sponsor and NC beforehand.
10. Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
11. Patients who are depending on the sponsor/CRO or investigational site as well as on the investigator.
12. Pregnancy or lactation period, or planning to become pregnant within 7 months after the end of treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (21):
- Germany (21):
  - Universitätsklinikum Aachen, Aachen
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Praxis Krebsheilkunde für Frauen, Berlin
  - Medizinisches Zentrum Bonn Friedensplatz, Bonn
  - Universitätsklinikum Brandenburg an der Havel, Brandenburg
  - Studien GbR Braunschweig, Braunschweig
  - Städtisches Klinikum Dessau, Dessau
  - Frauenklinik Carl Gustav Carus, Dresden
  - Onkologische Schwerpunktpraxis, Dresden
  - Krankenhaus Nordwest gGmbH, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - ZAGO am Helios Klinikum Krefeld, Krefeld
  - Universitätsfrauenklinik Leipzig, Leipzig
  - Universitätsklinik der Johannes Gutenberg-Universität Mainz, Mainz
  - Ruppiner Kliniken GmbH, Neuruppin
  - Sana Klinikum Offenbach, Offenbach
  - Klinikum Südstadt Rostock, Rostock
  - Caritas Klinikum St. Theresia, Saarbrücken
  - Krankenhaus Saarlouis vom DRK, Saarlouis
  - Christliches Klinikum Unna gGmbH, Unna

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period:01.02.2018 - 28.03.2023
Pre-assignment Details: A total of 204 patients were planned to be randomized. Due to slow recruitment of the trial, the recruitment was prematurely terminated after randomization of the 89th patient.
Groups:
- Arm B: * Carboplatin/PLD
  * Carboplatin/Gemcitabine
  * Carboplatin/Paclitaxel Patients will be treated for 6 cycles or until PD, unacceptable toxicity or patient's wish to discontinue, whichever occurs first.
  Trabectidin (Yondelis): To compare QoL in patients treated with trabectedin/PLD vs. other standard combination therapy of carboplatin/ PLD, carboplatin/ gemcitabine, or carboplatin/ paclitaxel
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 45 | 44
Completed | 44 | 41
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.9) | 64.9 (9.6) | 62.5 (10.5)
Age, Customized [Count of Participants; unit: Participants]
  < 70 years | 36 | 27 | 63
  >= 70 years | 8 | 14 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — The formula is BMI = kg/m²; (kg = person's weight in kilograms; m² =height in metres squared)
  kg/m² | 25.3 (5.2) | 26.2 (5.5) | 25.7 (5.4)
ECOG [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all predisease performance without restriction;
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work;
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours;
  3. - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours;
  4. - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair;
  5. - Dead
  Participants
    0 | 17 | 13 | 30
    1 | 27 | 27 | 54
    2 | 0 | 1 | 1
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
Localization of the primary tumor [Number; unit: participants]
  Primary peritoneal carcinoma | 3 | 4 | 7
  Primary ovarian carcinoma | 37 | 34 | 71
  Tube carcinoma | 4 | 3 | 7
Histology of primary tumor [Number; unit: participants]
  Clear cell | 2 | 3 | 5
  Mucinous | 0 | 1 | 1
  Serous | 42 | 37 | 79
Histological grade [Number; unit: participants] — grade 1 - well differentiated; grade 2 - moderately differentiated; grade 3 - poorly differentiated; grade 4 - undifferentiated; Lower grade tumours generally grow more slowly and are less likely to spread and metastasize than higher grade tumours.
  participants
    grade 1 | 2 | 0 | 2
    grade 2 | 1 | 1 | 2
    grade 3 | 6 | 2 | 8
    grade 4 | 0 | 0 | 0
    Missing | 35 | 38 | 73
Metastasis staging (according to TNM staging system) [Number; unit: participants] — M0 - no distant metastasis; M1 - distant metastasis (excluding peritoneal metastasis)
  participants
    M0 | 23 | 18 | 41
    M1 | 20 | 23 | 43
    Missing | 1 | 0 | 1
Number of previous chemotherapies [Number; unit: participants]
  1 | 32 | 36 | 68
  2 | 10 | 2 | 12
  3 | 1 | 3 | 4
  7 | 1 | 0 | 1
Number of relapses after previous therapy [Number; unit: participants]
  1 | 32 | 35 | 67
  2 | 9 | 3 | 12
  3 | 2 | 3 | 5
  7 | 1 | 0 | 1
Patient received at least one maintenance therapy with PARPi [Number; unit: participants] | 10 | 4 | 14
BRCA mutation [Number; unit: participants]
  YES | 5 | 4 | 9
  NO | 15 | 17 | 32
  Missing | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Difference in Quality of Life (QoL)
Description: The difference in QoL is defined as change of the mean score of the Trial Outcome Index (TOI) from baseline (TOI at randomization) compared to end of treatment (TOI at EOT) and is calculated as follows:
  Difference TOI = TOI at EOT - TOI at baseline.
  1. equals to 0 meaning no change in quality of life at EOT compared to baseline
  2. >0 meaning a detoriated quality of life at EOT compared to baseline. (The higher the number, the higher the detoriation.)
  3. <0 meaning an improved quality of life at EOT compared to baseline. (The lower the number, the higher the improvement.)
  TOI is calculated as mean of subscores concerning functional scales (e.g. physical function) and symptomal scales (e.g. body image, chemotherapy side effects, attitude to disease/treatment). Scores of each scale are transformed and ranges between 0-100. High scores for functional scales and symptomal scales meaning a low level of functioning and a high level of symptomatology/problems, respectively.
Time Frame: 12 month (from baseline to end of treatment)
Population: Five patients were excluded from the PP (per protocol) population due to violation of inclusion criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 42 | 38
units on a scale
  TOI at randomization (baseline) | 31.1 (15.6) | 28.7 (14.7)
  TOI at EOT | 36.9 (18.1) | 34.4 (16.6)
  Difference TOI: randomization over EOT | 6.5 (12.8) | 5.5 (12.7)

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as time (months) from randomization until date of the first occurrence of progression or recurrence, as determined by the investigator using CT criteria, or death from any cause.
Time Frame: 18 month
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 44 | 41
months | 8.2 [5.8 to 11.2] | 11 [9.0 to 13.6]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from randomization until date of death to any cause.
Time Frame: through study completion, up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 44 | 41
months | 14.9 [10.4 to 35.2] | 19.9 [11.2 to 30.7]

ADVERSE EVENTS:
Time Frame: through study completion, up to 3 years
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 40/44 | 38/41
Serious Adverse Events (participants affected / at risk) | 20/44 | 17/41
Other Adverse Events (participants affected / at risk) | 40/44 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=44) | Arm B (N=41)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 | 2
Ascites (General disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 1
Sepsis (General disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 4 | 2
Platelet count decrease (Blood and lymphatic system disorders) | 2 | 2
Worsening of general condition (General disorders) | 2 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Thromboembolic event (General disorders) | 0 | 1
g-GT increased (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Abdominal pain (General disorders) | 0 | 1
Anemia grade 2 (Blood and lymphatic system disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Hematoma (General disorders) | 1 | 0
Poor general condition (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=44) | Arm B (N=41)
Hypokalemia (Blood and lymphatic system disorders) | 4 | 0
Myalgia (General disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 10 | 6
Weight loss (General disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 11
Insomnia (General disorders) | 5 | 8
Hot flashes (General disorders) | 3 | 7
Stomach pain (General disorders) | 0 | 2
Dry skin (General disorders) | 3 | 4

LIMITATIONS AND CAVEATS:
Due to slow recruitment of the trial, the recruitment was prematurely terminated after randomization of the 89th patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT03164980/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03164980/SAP_001.pdf